CLINICAL TRIAL: NCT03532386
Title: Outcomes of Intra-Cytoplasmic Sperm Injection in Infertile Men With Non-tense Vaginal Hydrocele
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Lecturer, Tanta University
Other Study IDs: Ayman Shehata; Salah A Naglah (Other: Tanta University)
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Infertility, Male
Keywords: Infertility; male factor infertility; oligoasthenospermia; vaginal hydrocele
MeSH Terms: conditions — Infertility, Male; Infertility; Testicular Hydrocele | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group: Infertile men with oligoasthenospermia with non-tense vaginal hydrocele subjected to ICSI
  Interventions: Procedure: ICSI
- Control group: infertile men with oligoasthenospermia without hydrocele subjected to ICSI
  Interventions: Procedure: ICSI

INTERVENTIONS:
Procedure: ICSI — ICSI for both couples

SUMMARY:
Infertile men due to oligoasthenospermia with non-tense hydroceles are subjected to ICSI

DETAILED DESCRIPTION:
Sixty male infertile patients with Oligoasthenospermia were recruited from outpatient clinic of Urology Department, Tanta University. Patients were selected according to inclusion and exclusion criteria. The inclusion criteria were: (a) infertile couples due to male factor (b) Oligoasthenospermia (c) Normal hormonal profile (serum free and total testosterone, prolactin, Estrogen and LH), (d) presence or absence of non-tense vaginal hydrocel. The exclusion criteria were: (a) Presence of varicocele, (b) History of recent testicular trauma, (c) History of recent or old testicular inflammation, (d) Tense vaginal hydrocele and (e) presence of potential female pathologies.

Sample size calculation: With H0 denoting higher success rates for ICSI in absence of non-tense hydrocele and confidence level of 95% and interval of 5 the sample size was 30. The program used was Epi info 0.7.

Randomization and allocation: Enrolled patients were randomly allocated into 2 groups. The first group (n=30) who have oligoasthenospermia with non-tense vaginal hydrocele (Study group) and the second group (n=30) who have oligoasthenospermia with no hydrocele group (Control group). Randomization was done by computer-generated serial numbers where each number was enveloped. Each number denotes a certain allocation group. Allocation was by alternate method and envelope opening did not change allocation.

Methods: Males were assessed by genital examination, ultrasound and scrotal Doppler. Female partners were given long agonist stimulation protocols, Ovum pickup fertilization by sperms and then embryo transfer on day 5. Demographic data of both couples, duration of infertility, seminal parameters (WHO-2010) and results of ICSI in these couples were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Infertile couples due to male factor
* Oligoasthenospermia
* Normal hormonal profile (serum free and total testosterone, prolactin, Estrogen and LH)
* Presence or absence of non-tense vaginal hydrocele

Exclusion Criteria:

* Presence of varicocele
* History of recent testicular trauma
* History of recent or old testicular inflammation
* Tense vaginal hydrocele
* Presence of potential female pathology

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All infertile couples with male factor (oligoasthenospermia) due to non-tense hydrocele
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 2 weeks after ICSI
  Success of ICSI with positive pregnancy test in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Ayman Shehata Dawood, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: No
Not accepted to share patient data only results of study to be published